CLINICAL TRIAL: NCT01613001
Title: Obesity as a Risk Factor for Musculoskeletal Diseases in the U.S. Air Force: Associations and Implications for Force Readiness
Status: Completed | Type: Observational
Sponsor: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Responsible Party: Principal Investigator, Paul Crawford, Clinical Research Coordinator, Mike O'Callaghan Military Hospital
Other Study IDs: FWH20120036H
Record Dates: First submitted 2012-06-04; First posted 2012-06-06 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2013-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- DoD Beneficiaries: Exclusion: Active Duty Air Force members with the following conditions will be excluded from the study:
  * Documented preexisting musculoskeletal injury/disease before onset of obesity
  * Hypothyroidism/Hyperthyroidism
  * Hyperparathyroidism
  * Osteopenia/Osteoporosis
  * Nicotine dependence
  * Alcohol dependence
  * Eating disorders (anorexia nervosa, bulimia nervosa)
  * Cancer requiring chemotherapy or radiation therapy
  * Status-post gastrectomy
  * Status-post bilateral oophorectomy
  * Crohn's Disease
  * Ulcerative Colitis
  * Celiac Disease
  * Cushing's Disease
  * Prior to or during the study period, more than 6 months of taking proton pump inhibitors, medroxyprogesterone acetate, bisphosphonates, methotrexate, selective serotonin reuptake inhibitors, or inhaled/intranasal corticosteroids
  * Prior to or during the study period, more than 1 month of taking fluoroquinolones, oral or intramuscular corticosteroids, oral or intramuscular testosterone, or leuprolide

SUMMARY:
To study the first hypothesis, a retrospective cohort analysis of Air Force members from January 2005 to December 2010 will be performed to evaluate the association of obesity as an independent predictor variable with musculoskeletal disease as the dependent variable.

DETAILED DESCRIPTION:
To study the first hypothesis, a retrospective cohort analysis of Air Force members from January 2005 to December 2010 will be performed to evaluate the association of obesity as an independent predictor variable with musculoskeletal disease as the dependent variable. A second analysis will be performed on the same cohort using musculoskeletal disease as an independent predictor variable, as well as evaluating a potential interaction between obesity and musculoskeletal disease, to determine the association of these variables with the dependent variable of service member readiness for duty. The independent variables for the analyses include:

* Age
* Sex
* BMI
* Fitness data (PIMR: PFT scores, weight, height, BMI, abdominal circumference)
* Profile data (PIMR: Number of profiles, number of profiles due to musculoskeletal diagnoses, total days on duty limitation, total days on mobility limitation)
* Total number of deployments served
* All new musculoskeletal diagnoses (see attached abbreviated ICD-9 list)
* Incidence of member separation from AF
* Incidence of disability retirement
* X-rays
* Surgeries (orthopaedic, general)
* Referrals to the Orthopaedic Department
* Referrals to the Pain Clinic
* New diagnosis of diabetes mellitus
* Death

All data will be gathered by SG6H, Healthcare Informatics Division, and de-identified. Then the de-identified data will be coded and sent to the Principal Investigator for analysis. All informational data sets will be totally de-identified prior to releasing to the Principle Investigator to be analyzed by a statistician.

ELIGIBILITY:
Exclusion: Active Duty Air Force members with the following conditions will be excluded from the study:

* Documented preexisting musculoskeletal injury/disease before onset of obesity
* Hypothyroidism/Hyperthyroidism
* Hyperparathyroidism
* Osteopenia/Osteoporosis
* Nicotine dependence
* Alcohol dependence
* Eating disorders (anorexia nervosa, bulimia nervosa)
* Cancer requiring chemotherapy or radiation therapy
* Status-post gastrectomy
* Status-post bilateral oophorectomy
* Crohn's Disease
* Ulcerative Colitis
* Celiac Disease
* Cushing's Disease
* Prior to or during the study period, more than 6 months of taking proton pump inhibitors, medroxyprogesterone acetate, bisphosphonates, methotrexate, selective serotonin reuptake inhibitors, or inhaled/intranasal corticosteroids
* Prior to or during the study period, more than 1 month of taking fluoroquinolones, oral or intramuscular corticosteroids, oral or intramuscular testosterone, or leuprolide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: DoD Beneficiaries
Sampling Method: Non-Probability Sample
Enrollment: 67904 (Actual)
Dates: Start 2012-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Obesity vs musculoskeletal disease risk | within 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel Nye, MD, Principal Investigator — Mike O'Callaghan Military Hospital